CLINICAL TRIAL: NCT02931994
Title: Comparative Evaluation of the Plaque Removal Efficacy and Patient Acceptability of the Knotted Floss Technique With Conventional Flossing Technique in Type I Gingival Embrasures
Brief Title: Evaluation of Plaque Removal Efficacy and Patient Acceptability of Knotted Floss Technique in Type I Gingival Embrasures
Acronym: Knotfloss-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uttaranchal Dental & Medical Research Institute (Other)
Responsible Party: Principal Investigator, Aaron Gomes, Prof & Head, Dept of Periodontics & Oral Implantology, Uttaranchal Dental & Medical Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UttaranchalDMRI; UTN U1111-1188-4175 (Other: World Health Organization)
Record Dates: First submitted 2016-10-06; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Complication of Personal Oral Hygiene
Keywords: dental floss; gingival embrasure; oral hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A Phase 1 (No Intervention): 50% of sample are randomly assigned to Group A and are to utilise conventional flossing technique in the first phase of 6-weeks
- Group B Phase 1 (Active Comparator): 50% of sample are randomly assigned to Group B and are to utilise knotted floss technique in the phase 1 of 6-weeks
  Interventions: Other: Knotted floss technique
- Group A Phase 2 (Active Comparator): After a washout period of 2 weeks, those from Group A will use the knotted floss technique for a period of 6 weeks.
  Interventions: Other: Knotted floss technique
- Group B Phase 2 (No Intervention): After a washout period of 2 weeks, those from Group B will use the conventional floss technique for a period of 6 weeks.

INTERVENTIONS:
Other: Knotted floss technique — The subjects use the knotted floss technique. In this modification of conventional flossing technique, a knot is tied in the floss at any distance in the middle third of the floss length. The floss is inserted past the interdental contact point by the conventional finger flossing technique in the non-knotted area and then during the 'to and fro movement' on the tooth surface cervical to contact point, the knotted area is engaged through the embrasure (Gomes et al 2016)
  Arms: Group A Phase 2; Group B Phase 1

SUMMARY:
Removal and prevention of formation of dental plaque biofilms is one of the current hygiene regimen to prevent, reduce or even reverse the gingival and periodontal disease condition. In such endeavors of mechanical plaque removal, tooth-brushing and use of dental floss play an important role. Gomes et al have presented a modification in the use of knotted floss in wider embrasure areas. The modification in the dental floss has been done so as to increase the effective width of the floss. The purpose of this study is to compare the reduction of the clinical signs of plaque accumulation, gingival inflammation and gingival trauma in the area the knotted floss technique has been utilized versus the area where conventional flossing has been utilized in Type I gingival embrasures. Patients' acceptability of the knotted flossing technique will also be evaluated. This study is part of a larger study protocol involving different sample groups comparing the knotted floss technique with conventional dental flossing, use of interdental brushes and unitufted brushes in type II and type III embrasures as well.

DETAILED DESCRIPTION:
It has been well established that the origin of gingivitis and periodontal diseases occurs by the colonization, accumulation and subsequent maturation of bacterial plaque, (Loe et al 1965, Socransky 1970), and mediated by the host immunological response (Lewis et al, 2004). Since, oral bacteria in plaque biofilms are an essential component in the dental diseases processes, most of current preventive oral health care focuses on thorough plaque removal so as to prevent, reduce or even reverse the disease condition. (Suomi 1971, Schmid et al 1976). In such endeavors of thorough plaque removal and especially prevention of its further accumulation, dental surgeons and hygienists have commonly recommended daily mechanical plaque removal, specifically tooth-brushing. Use of toothbrush to mechanically remove plaque is extremely effective, but yet is not able to remove it thoroughly from interdental areas when used alone (Hansen & Gjermo 1971) Routine use of dental floss in conjunction with tooth-brushing has been shown to reduce the onset and severity of gingivitis (Bergenholtz & Britton 1980, Carter-Hanson et al 1996) Patients' reluctance and inability to perform flossing on a regular basis has been mentioned (Kresh 1976). In addition, to plaque control, patients also utilize flossing to clear the interdental areas wherein food impaction has occurred (Gjermo & Flotra 1970). Schmid (1984) has classified interdental embrasures, depending upon the filling of the gingival embrasure by the interdental papilla. Hence in Type I, floss is used, and in Type II and III the incrementally wider proxabrush and unitufted brush are used respectively. Gomes et al have presented a modification in the use of knotted floss in wider embrasure areas. (Gomes et al 2016). The modification in the dental floss had been done so as to increase the effective width of the floss. This enables it to be used in embrasures wider than that recommended for conventional floss. In this modification, a knot is tied in the floss at any distance in the middle third of the floss length. The floss is inserted past the interdental contact point by the conventional finger flossing technique in the non-knotted area and then during the 'to and fro movement' on the tooth surface cervical to contact point, the knotted area is engaged through the embrasure (Gomes et al 2016) The purpose of this study is to compare the reduction of the clinical signs of plaque accumulation, gingival inflammation and gingival trauma in the area the knotted floss technique has been utilized versus the area where conventional flossing has been utilized in Type I gingival embrasures. Patients' acceptability of the knotted flossing technique will also be evaluated. This study is part of a larger study protocol involving different sample groups comparing the knotted floss technique with conventional dental flossing, use of inter-dental brushes and unitufted brushes in type II and type III embrasures as well.

Study Design:

A sample size of thirty subjects will be selected based on the model used by Carter-Hanson et al 1996. Prior to commencement of the actual study, each volunteer will receive written and verbal instructions on the two techniques. The principal and third investigator will demonstrate to the volunteers both techniques on models, for half hour counseling session, for three consecutive days. Each counseling session will not have more than 10 participants. On the third day the volunteer's proficiency on models in both techniques will be confirmed by both demonstrators separately, informed consent will be taken and the volunteer will be enrolled as subject into the fourteen week, 2-phase crossover, single (examiner) blind study protocol with washout in-between phases. Failure by the volunteer to perform the techniques as instructed will result in another counseling session of half hour or he/she will not be included in the study protocol.

In the first phase, 50% of the subjects will be randomly assigned to use either conventional flossing technique, while the other 50% will be assigned to use the knotted floss technique. Only the first author know about which subject will be assigned to which technique. The treatment phase will consist of 6 weeks of daily use of the assigned technique followed by a 'washout period' of 14 days, following which will start the second treatment phase wherein the subject will use the other flossing technique. i.e those using the conventional flossing technique will now use the knotted flossing technique and vice versa. At the baseline appointment for each phase, every subject will be given their assigned floss products. Subjects that will be assigned to conventional flossing will receive ninety pieces of waxed floss, fifteen centimeters in length each piece, (Reach¬® by Johnson & Johnson Inc.) equally divided in three ziplock® bags. Subjects that will be assigned to knotted flossing technique will receive the same except that every floss thread will have a simple knot at around the middle. Each subject also will receive a sample of Colgate® Soft Toothbrush and Dentifrice (Colgate® Inc). The registered subjects will be instructed to brush their teeth twice a day in their customary manner using the above toothbrush and dentifrice provided and cautioned not to use any other oral hygiene aid except for the assigned floss twice a day. They will be instructed to wrap the floss around their middle or index finger and gently slide the floss between the teeth and move it along the gum margin, curved into "c" shape. After this, they will have to move the floss up and down several times between each tooth without using excessive pressure, finally allowing it out through embrasure. The subjects will have to return to the third author any unused floss products at the end of the phase. During the 'washout period' the subjects will be instructed to perform normal oral hygiene practices of tooth-brushing with dentifrice and refrain from using any floss or any additional plaque control aids. The "washout" period is designed so as to give subjects time to return to their original oral status and establish parity in baseline clinical measurements prior to starting the second treatment phase. Such a 'washout' in study design allowed use of 50% lesser subjects.

Clinical evaluations:

Clinical evaluations of all subjects will be done at 2-weekly intervals, namely baseline, 2 weeks, 4 weeks and 6 weeks of each treatment phase. Both adjacent teeth and gingiva at test sites will be scored for the Rustogi Modification of Navy Plaque Index, the Modified Gingival Index (Lobene 1986) and the Modified Papillary Bleeding Index (Barnett 1980). A plaque disclosing agent will be used to identify the location and amount of plaque. Additionally, gingival trauma will be assessed as presence or absence of signs of trauma in the marginal and papillary gingiva of adjacent teeth. The facial and lingual surfaces will be examined visually for gingival lacerations. Presence of laceration, floss cut, or demarcation line/indentation at the site will be scored as one, while a score of zero (0) will be recorded in the absence of any signs of trauma. The score per subject will be obtained by totaling all scores and dividing by number of sites examined (Carter-Hanson 1996).

The indices will be recorded by second and fourth investigator. Intra- and inter-examiner reliability will be established prior to commencement of the study and at two weekly intervals. The study schedule will be so distributed such that not more than six subjects report for examination on any given day of the week. The two examiners will have no knowledge as to which technique the subject is using and the amount of unused floss if any at end of phase.

Subject compliance A compliance diary will also be given to each subject at the baseline appointment of each treatment phase and will be collected at the end of each phase by third investigator. The subjects will be instructed to record each flossing experience in this diary and any other event he/she felt significant. Compliance will further be established by dispensing a specific amount (90 pieces) of assigned floss product per treatment phase. At the conclusion of each treatment phase, the subjects will return to principal or third investigator, any unused portion of floss product and thus non-compliance will be estimated. Additionally, the patient satisfaction questionnaire will substantiate subject compliance. This questionnaire will be answered by every subject at the end of the second and final phase.

ELIGIBILITY:
Inclusion Criteria:

* have one type I gingival embrasure in the premolar first molar area.
* full mouth Plaque Index score ≥1.8 (Silness and Loe 1964)
* full mouth Gingival Index ≥ 1.0 (Loe and Silness 1963)
* good general health,
* have all teeth present in quadrant being tested and opposing quadrant
* be available for a 14 week study period,
* be ready to abide with the study criteria,
* minimum education of grade 12

Exclusion Criteria:

* have used in previous 2months oral hygiene aids other than tooth-brushing like dental flossing, mouthwashes and water jet irrigating systems
* habit of unilateral mastication for ≥2 months,
* medical history of diabetes mellitus, hepatitis, pregnancy or requiring any antibiotic prophylaxis,
* having drug history in preceding two months of use of antibiotics, hormonal supplements, steroids, non steroidal anti-inflammatory medications, oral contraceptives or any drug that influence gingival tissue,
* taking part in any other clinical or drug trial including taking part in other study groups related to the evaluation of knotted floss technique,
* having physical handicap limiting the ability for oral hygiene and effective use of dental floss,
* had orthodontic treatment
* having gross dental caries
* having advanced periodontitis (more than one pocket ≥ 6mm),
* had active periodontal treatment like scaling, root planing, curettage, periodontal surgery in the previous 8weeks,
* had any adverse oral habit like smoking, tobacco chewing or habits of self gingival mutilation,
* had history of trauma or surgery to the jaws.
* teeth adjacent to the embrasure area selected are having proximal caries or gross occlusal caries, or having proximal restorations, crowns, onlays or inlays.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rustogi modification of Navy Plaque Index - 6weeks | 6 weeks
  Rustogi modification of Navy Plaque Index will be assessed at 6-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Lobene's Modified Gingival Index - 6weeks | 6 weeks
  Lobene's Modified Gingival Index will be assessed at 6-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Barnett's Modified Papillary Bleeding Index - 6weeks | 6 weeks
  Barnett's Modified Papillary Bleeding Index will be assessed at 6-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Gingival Trauma Index (as described by Carter-Hanson et al 1996)- 6weeks | 6 weeks
  Gingival Trauma will be assessed at 6-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2.
  The Gingival Trauma induced by improper flossing will be assessed by the technique described by Carter-Hanson et al 1996. All interdental areas of the facial and lingual surfaces of the gingiva will be examined for gingival lacerations and indentations, using a mouth mirror, light, and after gently air-drying the gingiva. A score of one (1) will be given to facial and lingual surface separately when floss trauma is identified as a demarcation line or laceration. A score of zero (0) will be recorded if no such trauma is present.
  The Gingival Trauma Index score per subject will be obtained by totalling all scores and dividing by number of sites examined.

SECONDARY OUTCOMES:
Rustogi modification of Navy Plaque Index - baseline | baseline
  Rustogi modification of Navy Plaque Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Lobene's Modified Gingival Index - baseline | baseline
  Lobene's Modified Gingival Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Barnett's Modified Papillary Bleeding Index - baseline | baseline
  Barnett's Modified Papillary Bleeding Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Gingival Trauma Index (as described by Carter-Hanson et al 1996) - baseline | baseline
  Gingival Trauma Index will be assessed at baseline for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2.
  The Gingival Trauma induced by improper flossing will be assessed by the technique described by Carter-Hanson et al 1996. All interdental areas of the facial and lingual surfaces of the gingiva will be examined for gingival lacerations and indentations, using a mouth mirror, light, and after gently air-drying the gingiva. A score of one (1) will be given to facial and lingual surface separately when floss trauma is identified as a demarcation line or laceration. A score of zero (0) will be recorded if no such trauma is present.
  The Gingival Trauma Index score per subject will be obtained by totalling all scores and dividing by number of sites examined.
Rustogi modification of Navy Plaque Index - 2 weeks | 2 weeks
  Rustogi modification of Navy Plaque Index will be assessed at 2 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Lobene's Modified Gingival Index - 2 weeks | 2 weeks
  Lobene's Modified Gingival Index will be assessed at 2 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Barnett's Modified Papillary Bleeding Index - 2 weeks | 2 weeks
  Barnett's Modified Papillary Bleeding Index will be assessed at 2 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Gingival Trauma Index (as described by Carter-Hanson et al 1996) - 2 weeks | 2 weeks
  Gingival Trauma Index will be assessed at 2-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2.
  The Gingival Trauma induced by improper flossing will be assessed by the technique described by Carter-Hanson et al 1996. All interdental areas of the facial and lingual surfaces of the gingiva will be examined for gingival lacerations and indentations, using a mouth mirror, light, and after gently air-drying the gingiva. A score of one (1) will be given to facial and lingual surface separately when floss trauma is identified as a demarcation line or laceration. A score of zero (0) will be recorded if no such trauma is present.
  The Gingival Trauma Index score per subject will be obtained by totalling all scores and dividing by number of sites examined.
Rustogi modification of Navy Plaque Index - 4 weeks | 4 weeks
  Rustogi modification of Navy Plaque Index will be assessed at 4 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Lobene's Modified Gingival Index - 4 weeks | 4 weeks
  Lobene's Modified Gingival Index will be assessed at 4 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Barnett's Modified Papillary Bleeding Index - 4 weeks | 4 weeks
  Barnett's Modified Papillary Bleeding Index will be assessed at 4 weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2
Gingival Trauma Index (as described by Carter-Hanson et al 1996) - 4 weeks | 4 weeks
  Gingival Trauma Index will be assessed at 4-weeks for all subjects in Group A Phase 1, Group B Phase 1, Group A Phase 2, and Group B Phase 2.
  The Gingival Trauma induced by improper flossing will be assessed by the technique described by Carter-Hanson et al 1996. All interdental areas of the facial and lingual surfaces of the gingiva will be examined for gingival lacerations and indentations, using a mouth mirror, light, and after gently air-drying the gingiva. A score of one (1) will be given to facial and lingual surface separately when floss trauma is identified as a demarcation line or laceration. A score of zero (0) will be recorded if no such trauma is present.
  The Gingival Trauma Index score per subject will be obtained by totalling all scores and dividing by number of sites examined.

OTHER OUTCOMES:
Patient satisfaction questionnaire | 14 weeks ( at end of study)
  Patients were asked to answer simple objective questionnaire selecting which technique was better with respect to ease of use, time taken for flossing, which technique was more painful and sensitive, which technique had better ability to clean, which technique they would prefer to continue in future?

CONTACTS AND LOCATIONS:
Overall Officials: Aaron F Gomes, MDS, Principal Investigator — Uttaranchal Dental and Medical Research Institute
Locations (1):
- Knotted Floss Study; Uttaranchal Dental and Medical Reserach Institute, Dehradun, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Background] Socransky SS. Relationship of bacteria to the etiology of periodontal disease. J Dent Res. 1970 Mar-Apr;49(2):203-22. doi: 10.1177/00220345700490020401. No abstract available. PMID 4313844
- [Background] Lewis MW, Holder-Ballard C, Selders RJ Jr, Scarbecz M, Johnson HG, Turner EW. Comparison of the use of a toothpick holder to dental floss in improvement of gingival health in humans. J Periodontol. 2004 Apr;75(4):551-6. doi: 10.1902/jop.2004.75.4.551. PMID 15152819
- [Background] Suomi JD. Prevention and control of periodontal disease. J Am Dent Assoc. 1971 Dec;83(6):1271-87. doi: 10.14219/jada.archive.1971.0471. No abstract available. PMID 4940401
- [Background] Schmid MO, Balmelli OP, Saxer UP. Plaque-removing effect of a toothbrush, dental floss, and a toothpick. J Clin Periodontol. 1976 Aug;3(3):157-65. doi: 10.1111/j.1600-051x.1976.tb01863.x. PMID 1067277
- [Background] Hansen F, Gjermo P. The plaque-removing effect of four toothbrushing methods. Scand J Dent Res. 1971;79(7):502-6. No abstract available. PMID 5289846
- [Background] Kresch CH. Finger-manipulated and floss-holder flossing: a comparison of the habit formation. Gen Dent. 1976 Jul-Aug;24(4):35. No abstract available. PMID 1065605
- [Background] Gjermo P, Flotra L. The effect of different methods of interdental cleaning. J Periodontal Res. 1970;5(3):230-6. doi: 10.1111/j.1600-0765.1970.tb00722.x. No abstract available. PMID 4254187
- [Background] Schmid M. Plaque control. In: Carranza F, editor. Glickmn's clinical periodontology. 6th ed. Philadelphia: W.B Saunders Company; 1984. p. 689-690
- [Background] Gomes A, Meru S, Rekhi A. Knotted floss technique. J Adv Res Dent Oral Health 2016;1(1):6-7
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Rustogi KN, Curtis JP, Volpe AR, Kemp JH, McCool JJ, Korn LR. Refinement of the Modified Navy Plaque Index to increase plaque scoring efficiency in gumline and interproximal tooth areas. J Clin Dent. 1992;3(Suppl C):C9-12. PMID 1306676
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Barnett M, Ciancio S. and Mather M. The modified papillary bleeding index: comparison with gingival index during the resolution of gingivitis. J Prev Dent 1980; 6:135-138
- [Result] Bergenholtz A, Brithon J. Plaque removal by dental floss or toothpicks. An intra-individual comparative study. J Clin Periodontol. 1980 Dec;7(6):516-24. doi: 10.1111/j.1600-051x.1980.tb02158.x. PMID 6938530
- [Result] Carter-Hanson C, Gadbury-Amyot C, Killoy W. Comparison of the plaque removal efficacy of a new flossing aid (Quik Floss) to finger flossing. J Clin Periodontol. 1996 Sep;23(9):873-8. doi: 10.1111/j.1600-051x.1996.tb00626.x. PMID 8891940
- [Result] Asadoorian J. Canadian dental hygienists association position statement on flossing. Can Jour Dent Hygienist. 2006;40(3):1-10
- [Result] Carr MP, Rice GL, Horton JE. Evaluation of floss types for interproximal plaque removal. Am J Dent. 2000 Aug;13(4):212-4. PMID 11763934